CLINICAL TRIAL: NCT02115607
Title: Quantitative Subharmonic Breast Imaging: Subharmonic Imaging and Pressure Estimation for Monitoring Neoadjuvant Chemotherapy
Brief Title: Subharmonic Imaging and Pressure Estimation for Monitoring Neoadjuvant Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13S.215; JT 2973 (Other: JeffTrial Number)
Record Dates: First submitted 2014-03-24; First posted 2014-04-16 (Estimated); Results first posted 2019-10-31 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Interstitial fluid pressure; Angiogenesis; Contrast enhanced ultrasound imaging; Subharmonic imaging; Subharmonic pressure estimation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Definity infusion (Experimental): Infusion of Definity (Perflutren Lipid Microspheres)
  Interventions: Drug: Definity infusion

INTERVENTIONS:
Drug: Definity infusion — 3 ml of Perflutren Lipid Microspheres (Definity) mixed in 50 ml of saline is infused at a rate of approximately 4ml/min
  Other Names: Perflutren Lipid Microspheres

SUMMARY:
This is a diagnostic accuracy study to evaluate if two novel ultrasound (US) techniques, quantitative 3D subharmonic imaging (SHI) and Subharmonic Aided Pressure Estimation (SHAPE), used with an intravenous ultrasound contrast agent (Definity, Lantheus Medical Imaging, Billerica, MA), can track changes in locally advanced breast cancer (LABC) angiogenesis and interstitial fluid pressure (IFP), respectively, by studying women undergoing neoadjuvant chemotherapy before as well as with around 10% and 60% (in part 1) or 30% (in part 2) of the neoadjuvant chemotherapy treatment delivered and after completion of the neoadjuvant chemotherapy treatment. Results will be compared to MRI and pathology.

ELIGIBILITY:
Inclusion Criteria:

* Females
* Be diagnosed with T1 or greater LABC, any N and M0.
* Be scheduled for neoadjuvant chemotherapy
* Be at least 21 years of age.
* Be medically stable.
* If a female of child-bearing potential, must have a negative pregnancy test.
* Have signed Informed Consent to participate in the study.

Exclusion Criteria:

* Males
* Females who are pregnant or nursing.
* Patients with other primary cancers requiring systemic treatment.
* Patients with any metastatic disease.
* Patients undergoing neoadjuvant endocrine therapy.
* Patients with known hypersensitivity or allergy to any component of Definity.
* Patients with cardiac shunts or congenital heart defects.
* Patients with unstable cardiopulmonary conditions or respiratory distress syndrome.
* Patients with uncontrollable emphysema, pulmonary vasculitis, pulmonary hypertension or a history of pulmonary emboli.
* Patients who have received any contrast medium (X-ray, MRI, CT or US) in the 24 hours prior to the research US exam.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-03; Primary Completion 2018-05-23 (Actual); Study Completion 2018-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flemming Forsberg, PhD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Definity Infusion
Started | 17
Completed | 16
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Definity Infusion
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Subharmonic Aided Pressure Estimation (SHAPE) After Treatment for Complete Responders
Description: To evaluate the ability of SHAPE, used with Definity, to track changes in interstitial fluid pressure (IFP) by studying women undergoing neoadjuvant chemotherapy before as well as with around 10% and 30% of the neoadjuvant chemotherapy treatment delivered and comparing results to MRI and pathology.
Time Frame: from baseline to completion of neoadjuvant chemotherapy, average of 6 months
Population: six participants were not counted in the data analysis. 2 due to technical issues, 2 withdrew due to worsening of underlying disease, and 2 stopped their nedoadjuvant chemotherapy treatment unexpectedly. Data presented below is for those who achieved Complete Response (CR)
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Definity Infusion
Number analyzed (Participants) | 6
dB
  10% completion of neoadjuvant chemotherapy for | 3.23 (1.41)
  30% completion of neoadjuvant chemotherapy | 1.67 (1.09)

2. Primary Outcome: Subharmonic Aided Pressure Estimation (SHAPE) After Treatment for Partial Responders
Description: To evaluate the ability of SHAPE, used with Definity, to track changes in interstititial fluid (IFP) by studying women undergoing neoadjuvant chemotherapy before as well as with around 10% 30% of the neoadjuvant chemotherapy treatment delivered and after completion of the neoadjuvant chemotherapy treatment and comparing results to MRI and pathology.
Time Frame: from baseline to completion of neoadjuvant chemotherapy
Population: six participants were not counted in the data analysis. 2 due to technical issues, 2 withdrew due to worsening of underlying disease, and 2 stopped their nedoadjuvant chemotherapy treatment unexpectedly. Data presented below is for those who achieved Partial Response (PR)
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Definity Infusion
Number analyzed (Participants) | 5
dB
  10% completion of neoadjuvant chemotherapy for | -0.88 (1.46)
  30% completion of neoadjuvant chemotherapy | 0.06 (0.90)

3. Secondary Outcome: Subharmonic Imaging (SHI) Depiction of Breast Cancer Angiogenesis for Complete Responders
Description: To compare the 3D Subharmonic imaging (SHI) depiction of breast cancer angiogenesis in humans to CD31, an immunohistochemical predictor of angiogenesis.
Time Frame: From baseline to after surgery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Definity Infusion
Number analyzed (Participants) | 6
dB | 1.1 (1.9)

4. Secondary Outcome: SHI Depiction of Breast Cancer Angiogenesis for Partial Responders
Description: To compare the 3D SHI depiction of breast cancer angiogenesis in humans to CD31, an immunohistochemical predictor of angiogenesis.
Time Frame: After surgery; on average 6 months
Population: Data presented below is for those who achieved Partial Response (PR)
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Definity Infusion
Number analyzed (Participants) | 5
dB | 0 (1.2)

ADVERSE EVENTS:
Time Frame: Up to 1 hour post infusion of contrast agent
Arm/Group | Definity Infusion
All-Cause Mortality (participants affected / at risk) | 3/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-02-20): https://cdn.clinicaltrials.gov/large-docs/07/NCT02115607/Prot_SAP_000.pdf